CLINICAL TRIAL: NCT02260310
Title: The Effect of Acupuncture Protocol Involving in Weizhong (BL4) and Huantiao (GB30) Points in Treating Ankylosing Spondylitis
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Chengdu PLA General Hospital (Other)
Responsible Party: Principal Investigator, Yang Min, Ph.D, Chengdu PLA General Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: BL40GB30
Record Dates: First submitted 2014-10-03; First posted 2014-10-09 (Estimated); Last update posted 2017-04-04 (Actual); Status verified 2017-03

CONDITIONS: Ankylosing Spondylitis
MeSH Terms: conditions — Spondylitis, Ankylosing

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Weizhong and Huantiao (Experimental): Patients with Ankylosing Spondylitis use the Acupuncture Protocol Involving in Weizhong (BL4) and Huantiao (GB30) Points
  Interventions: Other: Weizhong and Huantiao
- A-shi point (Active Comparator): Patients with Ankylosing Spondylitis use the Acupuncture Protocol Involving in A-shi points, without including Weizhong (BL4) and Huantiao (GB30) Points
  Interventions: Other: A-shi point

INTERVENTIONS:
Other: Weizhong and Huantiao
  Arms: Weizhong and Huantiao
Other: A-shi point
  Arms: A-shi point

SUMMARY:
The purpose of this study is to evaluate the effect of acupuncture protocol involving in Weizhong (BL4) and Huantiao (GB30) points in treating ankylosing spondylitis.

ELIGIBILITY:
Inclusion Criteria:

* Eligible adult (≥18 years of age) patients
* had a diagnosis of AS for at least 3 months defined as definite by the 1984 modified New York criteria
* Eligible patients also had a Bath Ankylosing Spondylitis Disease Activity Index (BASDAI) of ≥4 (0-10 cm scale)
* A visual analogue scale (VAS) score for total back pain of ≥4 (0-10 cm scale)

Exclusion Criteria:

* Had received prior Acupuncture therapy
* With complete ankylosis of the spine, defined as the presence of bridging syndesmophytes at all intervertebral levels of the cervical and lumbar spine on lateral view spinal radiographs

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2014-10; Primary Completion 2018-01 (Estimated); Study Completion 2018-01 (Estimated)

PRIMARY OUTCOMES:
Change from Baseline in McGill Pain Questionnaire (MPQ) at 12 weeks | At 0 week, 6 weeks, 12 weeks
Change from Baseline in Visual Analog Scale at 12 weeks | At 0 week, 6 weeks, 12 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- 270 Rongdu street, Jin-niu district,Rheumatology Center of Integrated Medicine, General Hospital of Chengdu Military Area Command PLA，, Chengdu, Sichuan, China